CLINICAL TRIAL: NCT07202273
Title: A Feasibility Study of Simulation-Free, Single-Fraction Palliative Radiation Therapy for Treatment of Bone Metastases (SIM-FREE RT)
Brief Title: Simulation-Free, Single-Fraction Palliative Radiation Therapy for Treatment of Bone Metastases
Acronym: SIM-FREE RT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI193478
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-09

CONDITIONS: Bone Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Simulation-free, single-fraction palliative radiation therapy (Experimental)
  Interventions: Radiation: simulation-free, single-fraction palliative radiation therapy

INTERVENTIONS:
Radiation: simulation-free, single-fraction palliative radiation therapy — Radiation will be delivered in a single fraction. The recommended prescription dose is 8 Gy with external beam radiation therapy.

SUMMARY:
The goal of this study is to provide proof that patients can be treated with simulation-free, single-fraction palliative radiation therapy with a single in-person visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years.
* Diagnosis of any cancer with one to two painful and treatable metastatic bone lesions.
* Bone metastases are causing pain or instability in the opinion of the treating investigator.
* Amenable to single fraction radiation therapy per the discretion of the treating physician.
* CT collected within 60 days of registration with adequate visualization of target site as determined by the treating investigator.
* ECOG Performance Status ≤ 2.
* Participants must adhere to the following sex and contraceptive/barrier requirements:

  * If participant is of childbearing potential, they must have a negative pregnancy test ≤ 14 days before the planned date of radiation therapy. This may be completed on the day of radiation if results from the pregnancy test are available for review before treatment.
  * For participants of non-child bearing potential: The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * < 50 years of age:

      * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
      * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution

        ---≥ 50 years of age:
      * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
      * Had radiation-induced menopause with last menses >1 year ago; or
      * Had chemotherapy-induced menopause with last menses >1 year ago
    * Participants of childbearing potential and participants with a sexual partner of childbearing potential must agree to use a highly effective method of contraception.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Evidence of spinal cord compression caused by the bone metastases to be treated.
* Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Medical, psychiatric, cognitive, or other conditions that may compromise the participant's ability to understand the participant information, give informed consent, comply with the study protocol or complete the study.
* Participants taking prohibited medications as described in Section 6.7.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
To assess the rate at which the intervention is delivered with fidelity to protocol. | 1 day
  To provide proof-of-concept that patients can be treated with simulation-free, single-fraction palliative radiation therapy with only a single in-person visit to Huntsman Cancer Hospital (HCH). This will be defined as receiving simulation-free, single-fraction radiation therapy with documented real-time approval by the radiation oncologist, medical physicist, and radiation therapist that the treatment adequately covers the target without unreasonable or unsafe differences.

SECONDARY OUTCOMES:
The percentage of patients who experience an improved Functional Assessment of Cancer Therapy Quality of Life Measurement in patients with bone pain score at 30 days post-treatment compared to baseline. | 30 days
  To assess whether the percentage of patients who experience an improvement in patient-reported quality of life related to bone pain after simulation-free, single-fraction palliative radiation therapy is consistent with a historical standard of 70%. Improved will be defined as an increase in total FACT-BP score of ≥ 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States